CLINICAL TRIAL: NCT01521065
Title: A Multicenter, Open-label Study to Evaluate the Clinical and Economic Benefits of Low Voltage Stereotactic Radiotherapy in Subjects With Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration (AMD)
Brief Title: An Open-label Study to Evaluate the Clinical and Economic Benefits of I-Ray in Patients With Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Acronym: ENDEAVOUR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oraya Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS002
Record Dates: First submitted 2012-01-18; First posted 2012-01-30 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Age-Related Macular Degeneration; Wet Macular Degeneration; Macular Degeneration; Eye Diseases; Retinal Diseases
Keywords: AMD; Wet AMD
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Eye Diseases; Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 16 Gy IRay (Experimental): 16 Gy IRay + PRN Lucentis®
  Interventions: Device: IRay

INTERVENTIONS:
Device: IRay — Approved dose of Anti-VEGF injection given at Day 0 followed by treatment with 16 Gy dose of IRay up to 14 days later.

SUMMARY:
The purpose of this study is to confirm the clinical and economic benefits of IRay treatment with respect to the number of anti-VEGF injections and frequency of visits during the first year after treatment for patients with wet Age-related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
The objective of this study is to confirm the clinical and economic benefits of low voltage external beam radiotherapy with the IRay with respect to number of anti-VEGF injections and frequency of ophthalmic assessments during the one year interval following treatment in subjects with neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

* Must have neovascular AMD and have received an anti-VEGF injections within 1 month prior to entering the study, and have the need for further treatment with anti-VEGF therapy.
* Must have a total lesion size of <12 disc areas and a CNV lesion with the greatest linear dimension of <6 mm, but not greater than 3 mm from the center of the fovea to the furthest point on lesion perimeter.
* Must have provided informed consent, documented it in writing, and have been given a copy of the signed informed consent form.
* Must be willing and able to return for scheduled treatment and follow-up examinations for the 3-year duration of the study.
* Must be at least 50 years of age.
* Women must be post-menopausal ≥1 year or surgically sterilized.
* Must have best corrected visual acuity of greater than or equal to 24 letters in the study eye and at least 20 letters in the fellow eye (if both eyes meet all the study criteria, then the eye with the worst vision should be selected as the study eye).

Exclusion Criteria:

* Present with any implanted device, where the device labeling specifically contraindicates subjects undergoing x-rays.
* An axial length of <20 mm (because of limitations of the IRay device) or >26 mm (to exclude subjects with pathologic myopia).
* Evidence of diabetes or retinal findings consistent with diabetic retinopathy, or retinopathy for any cause.
* Prior or concurrent therapies in the study eye for age related macular degeneration (other than intravitreal anti-VEGF), including submacular surgery, subfoveal thermal laser photocoagulation (with or without photographic evidence), transpupillary thermotherapy (TTT) and ocular photodynamic therapy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Rate of anti-VEGF injections during the first 12 months | 12 Months

SECONDARY OUTCOMES:
Time to first Anti-VEGF injection | Up to Month 12
Change in mean best-corrected visual acuity in the treated eye at month 12 | Month 12
Visual Functioning Questionnaire - 25 (VFQ-25) | Baseline & Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Royal Eye Hospital, Manchester, United Kingdom